CLINICAL TRIAL: NCT05242406
Title: Investigation of the Effect of Expiratory Muscle Strength Training Applied at Different Intensities on Systemic Inflammation and Oxidative Stress in Patients With Moderate Obstructive Sleep Apnea Syndrome
Brief Title: Effect of EMST Systemic Inflammation and Oxidative Stress in Patients With Moderate OSAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahi Evren Chest and Cardiovascular Surgery Education and Research Hospital (Other)
Responsible Party: Principal Investigator, NUREL ERTURK, Principal Investigator, Ahi Evren Chest and Cardiovascular Surgery Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021/363
Record Dates: First submitted 2022-01-12; First posted 2022-02-16 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Obstructive Sleep Apnea; Oxidative Stress; Respiratory Muscle Training
Keywords: Obstructive Sleep Apnea; Oxidative Stress
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- H-EMST (Experimental): In 60% of the maximum expiratory pressure (MEP), 25 breaths a day, 7 days / week, a total of 12 weeks will be trained with a 1-minute rest cycle in 5 breaths.
  Patients will be invited to control every 2 weeks. MEP measurements will be repeated and the training value will be adjusted in 60% of the new measurement.
  Interventions: Other: Expiratory muscle trainig
- L-EMST (Experimental): At 30% of the maximum expiratory pressure (MEP), 25 breaths, 7 days / week, a total of 12 weeks will be trained once a day with a 1-minute rest cycle in 5 breaths.
  Patients will be invited to control every 2 weeks. MEP measurements will be repeated and the training value will be adjusted in 30% of the new measurement.
  Interventions: Other: Expiratory muscle trainig

INTERVENTIONS:
Other: Expiratory muscle trainig — This exercise will be used to strengthen forced expiratory muscles.

SUMMARY:
It was aimed to investigate the effect of expiratory muscle strength training (EMST) applied at different intensities on systemic inflammation and oxidative stress in patients with moderate obstructive sleep apnea syndrome (OSAS). In the study, 32 male patients diagnosed with moderate OSAS will be included in the study. Participants will then be divided into 2 groups by block randomization. In the three-blind planned study; the first group will receive high-intensity %60 maximum expiratory pressure (MEP) EMST training, and the second group will be given low-intensity 30% of MEP, EMST training for 12 weeks. Disease-related symptoms, disease severity apnea-hypopnea index (AHI), oxidative stress index (OSI) and systemic inflammation level, exercise capacity, respiratory muscle strength, sleep quality, daytime sleepiness, and fatigue severity will be evaluated before and after the study.

DETAILED DESCRIPTION:
Primary outcome measures are; disease severity, oxidative stress index and systemic inflammation.

Secondary outcome measurements are; disease-related symptoms, exercise capacity, respiratory muscle strength, sleep quality, daytime sleepiness, and severity of fatigue.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients diagnosed with moderate OSAS by polysomnography in the Sleep Center of Ahi Evren Thoracic and Cardiovascular Surgery Training and Research Hospital,
2. Those who are between 19-60 years old,
3. Stable general health status,
4. Volunteer to participate in the research,
5. Not using NIMV device,

5) Patients who do not have a mental problem that will prevent cooperation will be included.

Exclusion Criteria:

1. Female gender,
2. Having a previous stroke,
3. Having an overlap syndrome,
4. Having any neurological, psychological or cardiac disease,
5. Uncontrolled hypertension and high blood glucose levels,
6. Severe obstructive nasal disease,
7. History of previous oropharyngeal surgery
8. Having a body mass index of 40 kg/m2 or more,
9. Using drugs, alcohol, sedative and hypnotic drugs,
10. Having a cognitive problem

Ages: 19 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Disease severity | 2 days
  Polysomnography recordings will be taken especially sleep efficiency and apnea-hypopnea index (AHI). Higher sleep efficiency and lower AHI values shows that patient have better status and lower disease severity
Oxidative stress-1 | 5 days
  TAS:Venous blood sample will be taken from the forearms of the patients in a 5 mL gel biochemistry tube with serum separator between 8.00-11.00 in the morning after an overnight fast and will be analyzed with a colorimetric kit.
Systemic inflammation-1 | 5 days
  CRP:biochemistry laboratory will work on the Abbott Architect C4000 (USA) clinical chemistry autoanalyzer.
Systemic inflammation-2 | 5 days
  TNF-a:After an overnight fast, venous blood samples will be taken from the forearms of the patients in a 5 mL gel biochemistry tube with serum separator between 8.00-11.00 in the morning and analyzed with the ELISA kit.
Systemic inflammation-3 | 5 days
  IL10:After an overnight fast, venous blood samples will be taken from the forearms of the patients in a 5 mL gel biochemistry tube with serum separator between 8.00-11.00 in the morning and analyzed with the ELISA kit.
Systemic inflammation-4 | 5 days
  IL-6:After an overnight fast, venous blood samples will be taken from the forearms of the patients in a 5 mL gel biochemistry tube with serum separator between 8.00-11.00 in the morning and analyzed with the ELISA kit.
Oxidative stress-2 | 5 days
  TOS:Venous blood sample will be taken from the forearms of the patients in a 5 mL gel biochemistry tube with serum separator between 8.00-11.00 in the morning after an overnight fast and will be analyzed with a colorimetric kit.

SECONDARY OUTCOMES:
Exercise capacity | 2 days
  6 minute walking testing (6MWT):The primary outcome is the distance covered in meters or converted measure (such as feet) over 6 minutes. To measure functional aerobic capacity or general fitness, this test may be used in conjunction with VO2 testing.
Maximal inspiratory and expiratory muscle strength | 2 days
  Maximal inspiratory and expiratory muscle strength will be evaluated with mouth pressure device.
Daytime sleepiness | 2 days
  Epworth Sleepiness Scale . Minimum and maximum scores: 0-24. The higher Epworth Sleepiness Scale score means the higher that person's average sleep propensity in daily life , or their 'daytime sleepiness'
Fatigue severity. | 2 days
  Fatigue Severity Scale (FSS)Minimum and maximum scores: 0-7. FSS scores higher than 4 shows high intensity fatigue perception
Sleep quality | 2 days
  The Pittsburgh Sleep Quality Index (PSQI). Minimum and maximum scores: 0-21. Higher PSQI scores show worse sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Adem Çelik, MD, Study Chair — Trabzon Ahi Evren Thoracic and Cardiovascular Surgery Training and Research Hospital; Sevim Kahraman Yaman, MD, Study Chair — Trabzon Ahi Evren Thoracic and Cardiovascular Surgery Training and Research Hospital; Hüseyin Yaman, MD, Study Chair — Karadeniz Technical University; Nurel Erturk, MsC, Principal Investigator — Trabzon Ahi Evren Thoracic and Cardiovascular Surgery Training and Research Hospital; Ebru Çalık Kütükçü, PhD, Study Director — Hacettepe University
Locations (1):
- Trabzon Ahi Evren Thoracic and Cardiovascular Surgery Training and Research Hospital, Ortahi̇sar, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Erturk N, Celik A, Kahraman Yaman S, Yaman H, Unal F, Calik Kutukcu E. Expiratory muscle strength training reduces oxidative stress and systemic inflammation in men with obstructive sleep apnea syndrome: a double-blinded, randomized parallel trial. Sleep. 2024 Dec 11;47(12):zsae221. doi: 10.1093/sleep/zsae221. PMID 39297486